CLINICAL TRIAL: NCT07152002
Title: A Phase 1, Randomized, Placebo-Controlled, Single and Multiple Ascending Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY4064912 in Healthy Participants and Participants With Overweight or Obesity
Brief Title: A Study of LY4064912 in Healthy Participants and With Overweight or Obesity
Acronym: YHAA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 27192; J5L-MC-YHAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Overweight or Obesity; Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: LY4064912 (Cohorts 1-6) (Experimental): LY4064912 administered subcutaneously (SC)
  Interventions: Drug: LY4064912
- Part A: LY4064912 (Cohort 6a) (Experimental): LY4064912 administered intravenously (IV)
  Interventions: Drug: LY4064912
- Part A: Placebo (Placebo Comparator): Placebo administered SC and IV
  Interventions: Drug: Placebo
- Part B: LY4064912 (Cohorts 7-10) (Experimental): LY4064912 administered SC
  Interventions: Drug: LY4064912
- Part B: Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- Part C: LY4064912 (Cohort 11) (Experimental): LY4064912 administered SC
  Interventions: Drug: LY4064912
- Part C: Placebo (Experimental): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4064912 — Administered SC
  Arms: Part A: LY4064912 (Cohorts 1-6); Part B: LY4064912 (Cohorts 7-10); Part C: LY4064912 (Cohort 11)
Drug: LY4064912 — Administered IV
  Arms: Part A: LY4064912 (Cohort 6a)
Drug: Placebo — Administered SC
  Arms: Part A: Placebo; Part B: Placebo; Part C: Placebo
Drug: Placebo — Administered IV
  Arms: Part A: Placebo

SUMMARY:
The purpose of this study is to evaluate how well LY4064912 is tolerated and what side effects may occur in healthy participants and participants with overweight and obesity - global. The study drug will be administered either subcutaneously (SC) (under the skin) or infusion intravenously (IV) (into a vein in the arm).

Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body.

ELIGIBILITY:
Inclusion Criteria:

* Age is 21-65 years old at Singapore Sites
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring

Part A: Body Mass Index (BMI) within the range greater than or equal to 21 and less than 30 kilogram per square meter (kg/m²)

Part B: a BMI greater than or equal to 27 and less than 45 kg/m²

Part C: a BMI greater than or equal to 21 and less than 35 kg/m²

* Parts A and C: Participants must weigh 60 kilograms (kg) or more at screening
* Have had a less than 5% change in body weight for 3 months before screening
* Safety laboratory tests are within normal reference range

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Have history of diabetes (except gestational diabetes) or current diagnosis of diabetes (any form), or have HbA1c greater than or equal to 6.5% (48 millimole per mole (mmol/mol)) at screening
* Are individuals of childbearing potential (IOCBP).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Postdose to Approximately Week 27
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY4064912 | Predose Up to Day 78
  PK: AUC of LY4064912
PK: Maximum Concentration (Cmax) of LY4064912 | Predose Up to Day 78
  PK: Cmax of LY4064912
Change from Baseline in Body Weight | Baseline to Approximately Week 27
  Change from Baseline in Body Weight
Effects of LY4064912 on Renal Hemodynamics and Renal Function | Baseline Up to Day 31
  Glomerular Filtration Rate (GFR)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (2):
  - Collaborative Neuroscience Network - CNS, Los Alamitos, California
  - ICON Early Phase Services, San Antonio, Texas
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No